CLINICAL TRIAL: NCT07261709
Title: Trifluridine/Tipiracil Plus Fruquintinib vs. Trifluridine/Tipiracil Plus Bevacizumab in Refractory Metastatic Colorectal Cancer: A Randomized, Controlled, Open-Label, Non-Inferiority Trial
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Peng Jian-jun, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAS-FUR
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-10

CONDITIONS: Refractory Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Trifluridine; tipiracil; HMPL-013; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trifluridine/tipiracil plus fruquintinib (Experimental)
  Interventions: Drug: Trifluridine/tipiracil plus fruquintinib
- Trifluridine/tipiracil plus bevacizumab (Active Comparator)
  Interventions: Drug: trifluridine/tipiracil plus bevacizumab

INTERVENTIONS:
Drug: Trifluridine/tipiracil plus fruquintinib — Trifluridine/tipiracil 35 mg/m² orally twice daily on days 1-5 and 8-12, repeated every 4 weeks, plus fruquintinib 4 mg orally once daily for 3 weeks followed by 1 week off, repeated every 4 weeks.
  Arms: Trifluridine/tipiracil plus fruquintinib
Drug: trifluridine/tipiracil plus bevacizumab — Trifluridine/tipiracil 35 mg/m² orally twice daily on days 1-5 and 8-12, repeated every 4 weeks, plus bevacizumab 5 mg/kg intravenously on day 1 every 2 weeks.
  Arms: Trifluridine/tipiracil plus bevacizumab

SUMMARY:
This study is an investigator-initiated, prospective, multicenter, randomized, controlled, open-label, non-inferiority trial designed to evaluate the efficacy and safety of trifluridine/tipiracil plus fruquintinib versus trifluridine/tipiracil plus bevacizumab in the treatment of refractory metastatic colorectal cancer.

DETAILED DESCRIPTION:
A total of 236 patients will be enrolled in this investigator-initiated, prospective, multicenter, randomized, controlled, open-label, non-inferiority trial.

Experimental group:

Trifluridine/tipiracil 35 mg/m² orally twice daily on days 1-5 and 8-12, repeated every 4 weeks, plus fruquintinib 4 mg orally once daily for 3 weeks followed by 1 week off, repeated every 4 weeks.

Control group:

Trifluridine/tipiracil 35 mg/m² orally twice daily on days 1-5 and 8-12, repeated every 4 weeks, plus bevacizumab 5 mg/kg intravenously on day 1 every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. All study participants must sign the informed consent form before any study-related procedures are initiated.
2. Aged 18-75 years, both males and females.
3. Histologically confirmed unresectable colorectal cancer.
4. RAS status known (mutant or wild-type).
5. Progression or intolerance after at least two prior systemic regimens that must have contained fluoropyrimidine-, oxaliplatin-, and irinotecan-based chemotherapy plus anti-VEGF therapy and/or anti-EGFR therapy.
6. At least one measurable lesion per RECIST v1.1.
7. Able to swallow oral tablets or capsules.
8. Estimated life expectancy ≥ 12 weeks.
9. ECOG performance status 0-1.
10. Adequate major organ function (within 7 days before randomization):

    Absolute neutrophil count ≥ 1.5 × 10⁹/L Platelet count ≥ 75 × 10⁹/L Hemoglobin ≥ 90 g/L (no transfusion within 7 days) Creatinine clearance ≥ 60 mL/min (Cockcroft-Gault formula) Total bilirubin ≤ 1.5 × upper limit of normal (ULN) AST and ALT ≤ 2.5 × ULN (≤ 5 × ULN if liver metastases present) Urinalysis showing proteinuria ≤ 1+ or 24-h urine protein < 1 g INR or PT ≤ 1.5 × ULN (acceptable if on anticoagulation and PT within intended therapeutic range)
11. Women of child-bearing potential must have a negative serum pregnancy test within 7 days before randomization; all participants and their partners must agree to use highly effective contraception from screening through at least 6 months after the last dose of study medication.

Exclusion Criteria:

* 1.Prior treatment with trifluridine/tipiracil, fruquintinib, or any other VEGF-receptor tyrosine-kinase inhibitor (e.g., apatinib, regorafenib, anlotinib).

  2.Pregnant or lactating women, or women who may become pregnant during the study.

  3.Anti-cancer therapy given ≤ 4 weeks before randomization (or not yet completed).

  4.Clinically relevant non-haematological CTCAE grade ≥ 3 toxicity from prior anti-cancer therapy that has not resolved to ≤ grade 1 (except alopecia and skin pigmentation).

  5.Symptomatic central-nervous-system metastases, unstable neurological status, or requirement for an increased steroid dose to control CNS disease.

  6.Severe or uncontrolled acute or chronic active infection. 7.History of active or interstitial lung disease, pneumonitis, or pulmonary arterial hypertension.

  8.Clinically significant active hepatitis of any cause, including but not limited to hepatitis B or C.

  9.Known HIV-positive status. 10.Uncontrolled hypertension (systolic BP ≥ 150 mmHg and/or diastolic BP ≥ 100 mmHg), uncontrolled arrhythmia, or symptomatic arrhythmia.

  11.Arterial thrombo-embolic event ≤ 6 months before randomization, including cerebrovascular accident or myocardial infarction.

  12.Major surgery ≤ 4 weeks before randomization (surgical incision must be fully healed before study drug administration), not yet recovered from previous surgery, or major surgery anticipated during the study.

  13.Radiotherapy ≤ 2 weeks before randomization, except short-course palliative radiotherapy for symptom relief.

  14.Any other clinically significant medical condition that, in the investigator's opinion, would compromise patient safety or study integrity.

  15.Concurrent or previous malignancy within 5 years, except adequately treated basal-cell or squamous-cell carcinoma of the skin or carcinoma in situ of the cervix.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-10-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
PFS | Time from the date of randomization to the first occurrence of disease progression (as assessed by the investigator according to RECIST v1.1) or death, whichever occurs first,up to 2 years
  Progression-free Survival

SECONDARY OUTCOMES:
OS | Time from the date of randomization to death from any cause up to 3 years
  Overall Survival
ORR | from randomization up to progressive disease or EOT due to any cause, up to 2 years
  Objective Response Rate
DCR | from randomization up to progressive disease or EOT due to any cause, up to 2 years
  Disease Control Rate
Safety and tolerance | from first dose to within 30 days after the last dose
  Safety and tolerance evaluated by incidence, severity and outcomes of adverse events (AEs) and categorized by severity in accordance with the NCI CTC AE Version 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- the first affiliated hospital of Sun Yat-sen University, Guangzhou, Guangdong 510080, Guangzhou, Guangdong, China